CLINICAL TRIAL: NCT03283956
Title: Safety and Efficacy of dRug-ElutiNg beADs Trans-arterial chemoEmbolization for Hepatocellular Carcinoma in Taiwan (SERENADE-T)
Brief Title: Safety and Efficacy of dRug-ElutiNg beADs Trans-arterial chemoEmbolization for Hepatocellular Carcinoma in Taiwan
Acronym: SERENADE-T
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Cheng-Kung University Hospital (Other); Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201708028RINC
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Hepatocellular Carcinoma Non-resectable; Chemoembolization, Therapeutic
MeSH Terms: interventions — Medical Records

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient records: Medical records of all patients who underwent DC bead TACE.
  Interventions: Device: Patient records

INTERVENTIONS:
Device: Patient records — Retrospective analysis of medical records of all patients who underwent DC Bead TACE at National Taiwan University Hospital, National Cheng Kung University Hospital, and Taichung Veterans General Hospital from 2010-2017/7

SUMMARY:
To evaluate efficacy and safety profile of DC bead® TACE in patients with hepatocellular carcinoma in Taiwan.

DETAILED DESCRIPTION:
To evaluate efficacy and safety profile of DC bead TACE in patients with hepatocellular carcinoma in Taiwan.

This is a multi-center, retrospective, single arm study to explore safety and efficacy of DC bead TACE in hepatocellular carcinoma (HCC) in Taiwan

Retrospective analysis of medical records of all patients who underwent DC Bead TACE at National Taiwan University Hospital, National Cheng Kung University Hospital, and Taichung Veterans General Hospital from 2010-2017/7.

All statistical data were analyzed with SPSS software (SPSS, IBM North America, New York, NY, USA). Demographic and baseline lab data are presented by using descriptive statistics Student's t-test. Survival analysis will includes all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of HCC, according to the AASLD diagnosis criteria for HCC.
* Patient received DC bead TACE.

Exclusion Criteria:

* Patients with current any other cancer except non-melanomatous skin cancer.
* Infiltrative HCC
* Patients received ≥2 consecutive sessions of TACE (≥2 TACE at the same admission, no matter it is cTACE or DC bead TACE)
* Patients received DC bead TACE and simultaneously received other therapy, such as radiotherapy, sorafenib etc.
* Presence of collateral vessel pathways potentially endangering normal territories during embolization.
* Presence of arteries supplying the lesion not large enough to accept DC Bead® microspheres.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical records of all patients who underwent DC bead TACE at National Taiwan University Hospital, National Cheng Kung University Hospital, and Taichung Veterans General Hospital from 2010-2017/7
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-09-13 (Estimated); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety of the DC bead TACE | One year.
  Safety of the DC bead TACE is evaluated based on the incidence of Grade 3 and Grade 4 toxicities up to 8 weeks following the procedure according to National Cancer Institute's Common Terminology Criteria for adverse events (CTCAE Version 4.03).

SECONDARY OUTCOMES:
Tumor response | One year.
  Tumor response is assessed on triphase CT or contrast-enhanced MR study according to modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hung Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No